CLINICAL TRIAL: NCT04734496
Title: Evaluation of Mechanisms of Sarcopenia in Chronic Inflammatory Disease (Chronic Liver Disease, Inflammatory Bowel Disease and Inflammatory Arthritis) Pre and Post Standard of Care Intervention; an Observational Study
Brief Title: Evaluation of the Mechanisms of Sarcopenia in Chronic Inflammatory Disease: Protocol for a Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Birmingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Matthew Armstrong, Principal Investigator, University of Birmingham
Other Study IDs: RG 18-053; 238190 (Other: IRAS)
Record Dates: First submitted 2021-01-18; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Chronic Liver Disease; Rheumatoid Arthritis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammatory Bowel Diseases | interventions — Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Muscle biopsy for histology, proteomics and genotyping Blood for RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Chronic Liver Disease: Patients with end-stage liver disease. Standard of care treatment will be nutrition and exercise as per European Association Study of Liver nutrition guidelines.
  Interventions: Other: National Healthcare System Standard of care for each disease type (National Institute for Health and Care Excellence guidelines)
- Rheumatoid Arthritis/Psoriatic arthropathy: Patients requiring biological therapy due to ongoing inflammation (requiring anti-Tumour Necrosis Factor therapy) - i.e. standard of care - escalation in therapy
  Interventions: Other: National Healthcare System Standard of care for each disease type (National Institute for Health and Care Excellence guidelines)
- Inflammatory Bowel Disease: Patients with Crohns or Ulcerative Colitis with ongoing inflammation (requiring anti-Tumour Necrosis Factor therapy) - i.e. standard of care - escalation in therapy
  Interventions: Other: National Healthcare System Standard of care for each disease type (National Institute for Health and Care Excellence guidelines)
- Healthy volunteers (n=20): Healthy volunteers

INTERVENTIONS:
Other: National Healthcare System Standard of care for each disease type (National Institute for Health and Care Excellence guidelines) — National Healthcare System Standard of care for each disease type (National Institute for Health and Care Excellence guidelines)
  Groups: Chronic Liver Disease; Inflammatory Bowel Disease; Rheumatoid Arthritis/Psoriatic arthropathy

SUMMARY:
Prospective, observational study to assess sarcopenia across three chronic inflammatory diseases: chronic liver disease, Inflammatory Bowel Disease, Rheumatoid Arthritis both before and after therapeutic intervention (standard of care treatment i.e. nutrition/exercise; biologic for IBD etc).

DETAILED DESCRIPTION:
Introduction: Several chronic inflammatory diseases co-exist with and accelerate sarcopenia (reduction in muscle strength, quantity and quality) and negatively impact on both morbidity and mortality. There is limited research on the extent of sarcopenia in such conditions, how to accurately assess it and whether there are generic or disease specific mechanisms driving sarcopenia.

Methods: This prospective cohort study is unique; it provides a multi-modal approach to assess sarcopenia across three chronic inflammatory diseases: chronic liver disease, Inflammatory Bowel Disease, Rheumatoid Arthritis both before and after therapeutic intervention. A total of 170 patients will be recruited (50 with Chronic liver disease, 20 with non-cirrhotic nonalcoholic fatty liver disease, 50 with Inflammatory Bowel Disease and 50 with Rheumatoid Arthritis) and including a comparison cohort of n=20 age-sex matched healthy individuals.

Participants will undergo 4 assessments at defined time points; weeks 0, 2, 12 and 24, with blood tests to assess endocrine and inflammatory status; anthropometric (hand grip strength; mid-arm muscle circumference; triceps skinfold thickness); functional testing (short physical performance battery and isokinetic dynamometry); imaging ( ultrasound and Magnetic Resonance Imaging of the quadriceps), and vastus lateralis muscle biopsy. Physical activity and sleep will be monitored using actigraphy, and quality of life via questionnaires. Food diaries for nutritional intake analysis will be sampled between 0-2, 12 and 24 weeks. Stool and urine samples will be sampled for future microbiome and metabolomics analysis, respectively.

This study will identify mechanisms across the groups and within each cohort, to further target interventions to reduce sarcopenia in the future. This is the first study to use a multi modal assessment to characterise sarcopenia in chronic disease. The multi-modal assessment includes serological, anatomical, functional and histological analyses to evaluate the deep phenotyping of these patients. The observational study of small sample sizes will allow potential future targets for intervention.

ELIGIBILITY:
Inclusion Criteria:

1. A formal confirmed diagnosis of their underlying chronic inflammatory condition:

   1. Inflammatory bowel disease cohort patients will have endoscopic or radiological evidence.

      Some of the Chronic liver disease cohort will have had a liver biopsy, serological and radiological confirmation will be sufficient.
   2. RA cohort, clinical, serological and radiological confirmation will be sufficient.
   3. Biologic therapy naïve on recruitment or commencing a new biologic if in the IBD or IA cohort.
2. Adults aged ≥ 18 years
3. Able to confirm written consent to the study
4. Biologic therapy naïve on recruitment or commencing a new biologic if in the IBD or RA cohort Pre-existing or current use of immunosuppressant agents or Disease Modifying Antirheumatic Drugs (DMARDs) are acceptable in all cohorts.
5. Meeting ACR (American College of Rheumatology) /EULAR (European League Against Rheumatism) 2010 or ACR 1987 Criteria for rheumatoid arthritis and starting DMARD therapy.
6. Meeting criteria of an inflammatory arthritis as per the American College of Rheumatology
7. Meeting criteria of liver cirrhosis including all Child Pugh scores from A-C as per British Association for the Study of the Liver guidance.
8. Meeting criteria for Inflammatory bowel disease as per the British Society of Gastroenterology guidance.
9. For muscle biopsy sampling (does not preclude patients from participating if they do not meet the below criteria) INR ≤ 1.6 Platelet count > 30

Exclusion Criteria:

1. Refusal or lack capacity to give informed consent.
2. Currently enrolled in an interventional trial with active treatment for their chronic disease condition.
3. Previously undergone LT or biliary intervention in the Chronic liver disease cohort.
4. Underlying or active cancer.
5. Biliary intervention if Chronic liver disease
6. For Muscle biopsies only (able to continue in study):

   1. Obvious injury to both thighs.
   2. Active bleeding of site, pre-procedure,
   3. Abnormal observation parameters.
   4. Acute illness.
   5. INR > 1.6.
   6. Platelet count < 30.
   7. Anticoagulation which cannot be paused due to increased risk to pre-existing co-morbidity.
7. For undergoing an Magnetic resonance imaging (MRI)

   1. Pacemaker.
   2. Metal work inserted that is not MRI compatible or further information cannot be obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic liver disease patients will be selected from those who undergo assessment for liver transplantation . A Non-alcoholic fatty liver disease (NAFLD) subset will be screened and recruited from the NAFLD clinic. For Inflammatory bowel disease and Rheumatoid Arthritis, all patients commencing a new biologic treatment (via biologic clinic screening or biologic registry screening) will be screened prior to therapy commencement.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Sarcopenia (Muscle Area) using Magnetic Resonance Imaging | 6 months
  Vastus lateralis and rectus femoris muscle axial cross sectional assessment will be measured at 50% of femur length
Sarcopenia (Muscle Area) using ultrasound | 6 months
  Vastus lateralis and rectus femoris muscle axial cross sectional assessment will be measured at 50% of femur length.

SECONDARY OUTCOMES:
Quality of Life questionnaire | 6 month
  Short Form-36 health-related Quality of Life questionnaire (Quality Metric Health Outcomes Solutions, Lincoln, USA)
Muscle biopsy of the Vastus lateralis | 6 month
  Muscle structure using standardised haemotoxylin/eosin and immunohistochemistry
Leg (Quadricep/Hamstring) strength | 6 month
  Leg strength/power by Isokinetic Dynamometry - the patient will be asked to extend the leg as strong as possible and then to flex, for 5 repetitions
Handgrip strength | 6 month
  Both hands using handheld Dynamometer (North Coast Medical, Morgan Hill)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Lord, PhD, Study Chair — University of Birmingham
Locations (1):
- Institute of Inflammation and Ageing (IIA) University of Birmingham Research Laboratories, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quinlan JI, Nicholson T, Bell C, Dhaliwal A, Williams FR, Allen SL, Choudhary S, Rowlands AV, Elsharkawy AM, Armstrong MJ, Greig CA, Lord JM, Jones SW, Breen L. Increased quadriceps intermuscular adipose tissue in chronic liver disease is associated with an altered muscle transcriptome compared with healthy age matched controls. Geroscience. 2025 Nov 14. doi: 10.1007/s11357-025-01982-2. Online ahead of print. PMID 41239110
- [Derived] Dhaliwal A, Williams FR, Quinlan JI, Allen SL, Greig C, Filer A, Raza K, Ghosh S, Lavery GG, Newsome PN, Choudhary S, Breen L, Armstrong MJ, Elsharkawy AM, Lord JM. Evaluation of the mechanisms of sarcopenia in chronic inflammatory disease: protocol for a prospective cohort study. Skelet Muscle. 2021 Dec 11;11(1):27. doi: 10.1186/s13395-021-00282-5. PMID 34895316